CLINICAL TRIAL: NCT01673893
Title: ClearWay Rx Readmission Registry
Acronym: ClearWay
Status: Completed | Type: Observational
Sponsor: Cardiovascular Institute of the South Clinical Research Corporation (Other)
Responsible Party: Sponsor
Other Study IDs: K061680
Record Dates: First submitted 2012-08-24; First posted 2012-08-28 (Estimated); Results first posted 2018-09-24 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Acute Myocardial Infarction
Keywords: ClearWay; Glycoprotein; Primary Coronary Intervention; Abciximab; ST Elevation Myocardial Infarction; Non-ST Elevation Myocardial Infarction; Medicare; Medicaid; Registry; catheterization; readmission; Acute Coronary Syndrome; ClearwayRx Catheter
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ST elevation myocardial infarction: The registry will record the use of the ClearWay™ Rx catheter during the index procedure, and assess whether or not the patient was readmitted within 30 days, related to the index procedure.
  1st Group/Cohort - ST elevation myocardial infarction
  Interventions: Device: ClearWay™ Rx catheter
- Non-ST elevation myocardial infarction/ACS/UNSTABLE ANGINA: The registry will record the use of the ClearWay™ Rx catheter during the index procedure, and assess whether or not the patient was readmitted within 30 days, related to the index procedure.
  2nd Group/Cohort - Non-ST elevation myocardial infarction/ACS/Unstable Angina
  Interventions: Device: ClearWay™ Rx catheter

INTERVENTIONS:
Device: ClearWay™ Rx catheter

SUMMARY:
The purpose of this registry is to determine if delivery of weight adjusted, in a large dose with either Abcixmab or Eptifibitide through the ClearWay™ RX, in patients admitted for primary coronary intervention lowers readmission rate. This is done in comparison to the historical control of the Medicare/Medicaid readmission database. The registry will record the use of the product during the index procedure, and determine whether or not the patient was readmitted within 30 days, related to the index procedure.

DETAILED DESCRIPTION:
The primary goal of this registry is to prospectively assess if delivery of weight adjusted, bolus only with either abcixmab or eptifibitide through the ClearWay™ RX in patients admitted for primary PCI lowers readmission rate in comparison to the historical control of the Medicare/Medicaid readmission database. The registry will record the use of the product during the index procedure, and assess whether or not the patient was readmitted within 30 days, related to the index procedure.

The ClearWay™ RX Local Therapeutic Infusion Catheter is a micro-porous PTFE balloon catheter designed for the localized infusion of various diagnostic and therapeutic agents into the coronary and peripheral vasculature. The ClearWay™ RX creates a low pressure fluid layer that surrounds the balloon, allowing more effective delivery of a prescribed therapeutic agent, without excessive stress and uncontrollable mechanical disruption seen with more traditional elastomeric devices. In addition, the ClearWay™ RX is a low pressure irrigating balloon system and non-compliant balloon that limits the amount of mechanical stress on the vessel wall.

The objective of this prospective registry is to evaluate whether intracoronary (IC) delivery of Glycoprotein IIb/IIIa inhibitors (GP IIb/IIIa) during Primary Coronary Intervention (PCI) can reduce the likelihood of 30 day readmissions as a result of the original coronary intervention. Intracoronary delivery of GP IIb/IIa inhibitor Abciximab in ST Elevation Myocardial Infarction has shown to reduce myocardial infarct size, no reflow or slow flow, improve TIMI flow and Myocardial Blush Grade2,3. The ICE trial4 (N=376) compared IC delivery of GP IIb/IIa inhibitor Eptifibitide bolus only administration, bolus with maintenance infusion of Eptifibitide, to standard intravenous (IV) bolus with maintenance infusion. At 24 month follow up, the Major Adverse Coronary Events (MACE) rate was lower in the IC bolus only group (2.5%) versus IC bolus and maintenance infusion (5.8%), and IV bolus with maintenance infusion (10.8%). Further, target lesion revascularization, and readmission rates were significantly lower in the IC bolus only arm, (10.9% versus 16.8% and 28% respectively).

ELIGIBILITY:
Inclusion Criteria:

* Acute Coronary Syndrome (ST elevation myocardial infarction or Non ST elevation myocardial infarction) patients requiring the use of the ClearWay™ Rx local therapeutic infusion catheter for intracoronary delivery of GP IIb/IIIa inhibitor.

Exclusion Criteria:

* Patients not meeting the above inclusion criterion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients presenting with myocardial infarction
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2011-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nick Cavros, MD, Principal Investigator — Cardiovascular Institute of the South
Locations (1):
- Cardiovascular Institute of the South Clinical Research Corporation, Lafayette, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krumholz, et al. Circulation 2009; 2:407-413.
- [Background] Thiele, et al. Circulation 2008 Vol. 118
- [Background] Romagnoli E, Burzotta F, Trani C, Biondi-Zoccai GG, Giannico F, Crea F. Rationale for intracoronary administration of abciximab. J Thromb Thrombolysis. 2007 Feb;23(1):57-63. doi: 10.1007/s11239-006-9000-0. PMID 17160551
- [Background] Hassan, et al. American Heart Journal. Volume 154;2:345-351.
- [Background] Curtis JP, Schreiner G, Wang Y, Chen J, Spertus JA, Rumsfeld JS, Brindis RG, Krumholz HM. All-cause readmission and repeat revascularization after percutaneous coronary intervention in a cohort of medicare patients. J Am Coll Cardiol. 2009 Sep 1;54(10):903-7. doi: 10.1016/j.jacc.2009.04.076. PMID 19712799

RESULTS

PARTICIPANT FLOW:
Groups:
- Readmission Results: The registry will record the use of the ClearWay™ Rx catheter during the index procedure, and assess whether or not the patient was readmitted within 30 days, related to the index procedure.
  ClearWay™ Rx catheter
Period: Overall Study
Arm/Group | Readmission Results
Started | 59
Completed | 59
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- ST Elevation Myocardial Infarction: The registry will record the use of the ClearWay™ Rx catheter during the index procedure, and assess whether or not the patient was readmitted within 30 days, related to the index procedure.
  1st Group/Cohort - STEMI: ST elevation myocardial infarction
- Non ST Elevation Myocardial Infarction/ACS/UNSTABLE ANGINA: The registry will record the use of the ClearWay™ Rx catheter during the index procedure, and assess whether or not the patient was readmitted within 30 days, related to the index procedure.
  2nd Group/Cohort - NSTEMI: Non-ST elevation myocardial infarction/ACS/Unstable Angina
- Total: Total of all reporting groups
Arm/Group | ST Elevation Myocardial Infarction | Non ST Elevation Myocardial Infarction/ACS/UNSTABLE ANGINA | Total
Number analyzed (Participants) | 43 | 16 | 59
Age, Customized [Number; unit: years]
  <50 years | 6 | 1 | 7
  50 to 65 years | 24 | 8 | 32
  65 to 75 years | 9 | 6 | 15
  >= 75 Years | 4 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 36 | 13 | 49

OUTCOME MEASURES:

1. Primary Outcome: 30 Day Readmissions
Description: Collecting data for STEMI and NSTEMI patients for 30 day readmissions after the STEMI or NSTEMI with use of the clearway catheter during the procedure.
Time Frame: 30 Days
Population: The above documentation shows the number of readmissions within 30days of post PCI with 7 subjects. The number of cardiovascular Admissiosn within 30 days that were not preplanned or elective are 3. The number of subjects compliant with the dual anti platelet therapy consists of 59 subjects who completed the study.
Measure: Number; unit: participants
Groups:
- No. Re-admission Within 30-days Post Pci: No. of Re-admission within 30-days post pci
- No. of Cardiovascular Admissions Within 30-days: No. of Cardiovascular Admissions within 30-days: not preplanned, not elective
- No. of Patients Compliant With DAPT: No. of patients compliant with Dual Anti Platelet Therapy
Arm/Group | No. Re-admission Within 30-days Post Pci | No. of Cardiovascular Admissions Within 30-days | No. of Patients Compliant With DAPT
Number analyzed (Participants) | 59 | 59 | 59
participants | 7 | 3 | 59

ADVERSE EVENTS:
Description: Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed on 7 participants with re-admissions within 30 days post pci and 3 participants who had Cardiovascular Admissions within 30-days that were not preplanned or elective. Re-admissions were captured for data purposes only, not followed.
Groups:
- EG000: Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed on 7 participants with re-admissions within 30 days post pci and 3 participants who had Cardiovascular Admissions within 30-days that were not preplanned or elective. Re-admissions were captured for data purposes only, not followed.
Arm/Group | EG000
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less